CLINICAL TRIAL: NCT04371874
Title: The Standardized and Economical Mode for the Prevention and Management of Chronic Cardiovascular Diseases: Matrix System From Rural Shaanxi ( MATRIX ) Ⅰ
Brief Title: The Standardized Management of Hypertension in Rural Shaanxi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Hongyan Tian, vice director, First Affiliated Hospital Xi'an Jiaotong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GS610101-Ⅰ
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Hypertension
Keywords: hypertension management; rural areas; control rate
MeSH Terms: conditions — Hypertension | interventions — Hydrochlorothiazide; Captopril; Nitrendipine; Aspirin

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Control (No Intervention): Hypertension of patients in the control group was managed with the original protocol including lifestyle by doctors in village clinic.
- Treatment with Ten Dollars Project (TDP) (Experimental): Hypertension of patients in the TDP group were managed with the protocol of "Ten Dollars Project (TDP)" by doctors in village clinic.
  Interventions: Drug: Hydrochlorothiazide, Captopril, Nitrendipine, Aspirin

INTERVENTIONS:
Drug: Hydrochlorothiazide, Captopril, Nitrendipine, Aspirin — The participants were grouped into a control group and a TDP group. Hypertension of patients in the control group was managed with the original protocol by doctors in village clinics. Patients in the TDP group were supplied with the TDP treatment, for whom different levels of oral administration plans to patients without drugs treatment in original protocol were: G 0 and G I, nifedipine (20mg, bid) or captopril (25mg, tid), hydrochlorothiazide (12.5mg, bid) for patients who couldn't tolerate previous drugs; G II, nifedipine (20mg, bid) plus hydrochlorothiazide (12.5mg, bid), or captopril (25mg, tid) plus hydrochlorothiazide (12.5mg, bid ), triple therapy for patients whose blood pressure did not reach target BP; G III, three drugs combination. Patients with drugs treatments in the original protocol were changed to be treated with the above antihypertension medications which were uniformly supplied by the government.
  Other Names: medications were uniformly supplied by the Chinese government
  Arms: Treatment with Ten Dollars Project (TDP)

SUMMARY:
The purpose of the study is to build a prevention and management system of hypertension in rural Shaanxi, China, which tries to use the standardized and economical methods to improve the outcome of chronic cardiovascular diseases.

DETAILED DESCRIPTION:
Hypertension is common in China, but there are low rates of awareness (36.0%), treatment (22.9%) and control (5.7%) in the hypertension population of an estimated 200 million adults, a figure generated from the nationwide China Patient-Centered Evaluative Assessment of Cardiac Events (PEACE) Million Person Project (MPP) . Substantial health and economic burdens are caused by hypertension, and adequate control of blood pressure (BP) has been a national public health priority. In China, nearly half of population are living in rural areas , where lower treatment and control rates of hypertension compared with urban areas. Expenditure of antihypertension medications and insufficient professional ability of rural doctors were the major problems facing hypertension management in rural areas of China with backward economies.

Absence of affordable medications prescribed may be a major barrier to adherence to medications. The rural doctors with insufficient professional ability had not to provide standard management of hypertension. So, an effective, cheap and simple hypertension control strategy was urgently needed in underdeveloped rural areas.

My center has been devoted to the study of hypertension in economically backward rural areas of Shaanxi Province in Western China for decades. We provided a cheap and simple hypertension management plan suitable for these areas. Because the cost of the management was about $10 dollars per year, the plan was called the ten dollars project (TDP). The TDP included a management system and a cheap treatment plan. The management software for hypertension was designed to help rural doctors with poor professional medical ability standardly manage hypertension adhering to the guidelines. Of course, a more effective and affordable treatment costing about ten dollars a year is the core of this system. The aim of this study was to measure whether the TDP can effectively improve the control of hypertension in rural areas.

ELIGIBILITY:
Inclusion Criteria:

* primary hypertension;
* Age ≥ 18 years old;

Exclusion Criteria:

* Secondary hypertension;
* the acute onset of cardiovascular events within three months;
* severe liver disease (ALT increased 2-fold greater than creatinine 2.5mg/dl);
* Severe cardiomyopathy, congenital heart disease, rheumatic heart disease
* malignancies
* allergic to study drugs
* with clear contraindications on study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1210 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
the improvement of control rate of hypertension with low-cost in rural Shaanxi | Patients in the TDP group accepted protocol of TDP to manage hypertension and patients in the control group were managed by the original protocol for six months. Compare the change of control rate at baseline and the end of the sixth month.
  value whether the protocol of TDP could improve the control rate of hypertension in rural Shaanxi

CONTACTS AND LOCATIONS:
Overall Officials: Hongyan Tian, Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- the first affiliated hospital of Xi'an Jiaotong university, Xi'an, China